CLINICAL TRIAL: NCT04923945
Title: A Multi-center, Open-label, Phase IIIb Confirmatory Clinical Trial to Evaluate the Efficacy, Safety and Tolerability of Savolitinib in Treating Locally Advanced or Metastatic NSCLC Patients With MET Exon 14mutations
Brief Title: Savolitinib for Treating Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-504-00CH2
Record Dates: First submitted 2021-05-30; First posted 2021-06-11 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Non-small Cell Lung Cancer Metastatic
MeSH Terms: interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine

STUDY DESIGN:
Intervention Model Description: locally advanced or metastatic NSCLC patients with MET exon 14 mutations without EGFR, ALK and ROS1 sensitive mutations who had disease progression or intolerable toxicity after previous therapy with platinum-based chemotherapeutic regimen and are treatment-naïve to c-MET therapy OR who did not receive any drug therapy for advanced tumors previously.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Savolitinib (Experimental): NSCLC
  Interventions: Drug: Savolitinib

INTERVENTIONS:
Drug: Savolitinib — Patients meeting the study inclusion criteria will receive Savolitinib [Savolitinib 600 mg, po, once per day (QD) continuously in patients with baseline weight ≥50 kg, and Savolitinib 400 mg, po, QD in patients with baseline weight <50 kg] in 21 day treatment cycle, until disease progression, death, intolerable toxicity or other termination criteria as specified in the protocol, whichever occurs earliest. Or patient will receive Savolitinib [Savolitinib 300 mg, po, twice per day (BID) continuously in patients with baseline weight ≥50 kg, and Savolitinib 200 mg, po, BID in patients with baseline weight <50 kg] in 21 day treatment cycle, until disease progression, death, intolerable toxicity or other termination criteria as specified in the protocol, whichever occurs earliest.

SUMMARY:
Treating Non-small Cell Lung Cancer (NSCLC) Patients with MET exon 14mutations with Savolitinib

DETAILED DESCRIPTION:
This is a single-arm, multi-cohort, multi-center, open-label, phase IIIb clinical study. The objective is to evaluate the efficacy and safety of Savolitinib in the treatment of locally advanced or metastatic NSCLC patients with MET exon 14 mutations. The study involves a Screening Period, a Treatment Period and a Follow-up Period. There are 53 study sites initiated and enrolled 203 advanced or metastatic NSCLC patients with MET exon 14 mutations

ELIGIBILITY:
Inclusion Criteria:

1. Fully aware this study and signed the informed consent form in voluntary manner, and willing and able to comply with the study procedure;
2. Age ≥18 years;
3. Histologically diagnosed locally advanced or metastatic NSCLC with MET exon 14 mutation;
4. Cohort 1: disease progression or intolerable toxicity after previous therapy with platinum-based chemotherapeutic regimen (for the patients who have received platinum-based adjuvant chemotherapy/radiotherapy, neoadjuvant chemotherapy/radiotherapy previously or radical radiochemotherapy for progressive disease, if the disease progression occurred < 6 months after the end of the last therapy, the patient belongs to failure after the first-line therapy); Cohort 2: no any previous systematic antitumor therapy for advanced diseases; Cohort 3: no any previous systematic antitumor therapy for advanced diseases;
5. Having measurable lesions (in accordance with RECIST 1.1 criteria);
6. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1, or Karnofsky performance status ≥80;
7. Survival is expected to exceed 12 weeks;
8. Adequate functionality in bone marrow, liver, kidney
9. Able to take or swallow the drug orally.
10. Female patients of childbearing potential must agree to use effective contraceptive methods from screening period to 30 days after discontinuation of the study drug,The male patients whose sexual partners are women of childbearing age must use condom during sexual intercourse during the study and within 6 months after discontinuation of study drug;

Exclusion Criteria:

1. Having gene mutations sensitive to targeted drugs for EGFR, ALK and ROS1;
2. Previous anti-MET therapy (including but not limited to crizotinib, Onartuzumab, etc.)
3. Currently having other malignant tumors, or having other infiltrating malignant tumors in the past 5 years. Stage I malignant tumor after radical treatment for at least 3 years, except those considered by investigators to have small possibility of recurrence. Patients with radically treated carcinoma in situ (non-infiltrating) and skin cancer other than malignant melanoma can be enrolled;
4. Having received antitumor therapy (including chemotherapy, hormone therapy, biotherapy, immunotherapy or traditional Chinese medicine for antitumor indication) within 3 weeks prior to the start of study treatment, or having received treatment with small molecular tyrosine kinase inhibitors (e.g., EGFR-TKI) within 2 weeks prior to the start of study treatment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) evaluated by the Independent Review Committee (IRC) (RECIST 1.1 criteria) | through study completion, an average of 3 years
  To evaluate the efficacy of Savolitinib in the treatment of locally advanced or metastatic NSCLC patients with MET exon 14 mutations

SECONDARY OUTCOMES:
Progression-free survival (PFS) (RECIST 1.1 criteria) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  To evaluate the efficacy of Savolitinib in the treatment of locally advanced or metastatic NSCLC patients with MET exon 14 mutations
incidence of various adverse events (AE) | through study completion, an average of 3 years
  To evaluate the safety and tolerability of Savolitinib in the treatment of locally advanced or metastatic NSCLC patients with MET exon 14 mutations

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu Y, Guo Q, Zhang Y, Fang J, Zhong D, Liu B, Pan P, Lv D, Wu L, Zhao Y, Li J, Liu Z, Liu C, Su H, Fan Y, Zhang T, Liu A, Jin B, Wang Y, Zhou J, Zhang Z, Ran F, Song X, Shi M, Su W, Lu S; study group. Savolitinib in patients in China with locally advanced or metastatic treatment-naive non-small-cell lung cancer harbouring MET exon 14 skipping mutations: results from a single-arm, multicohort, multicentre, open-label, phase 3b confirmatory study. Lancet Respir Med. 2024 Dec;12(12):958-966. doi: 10.1016/S2213-2600(24)00211-X. Epub 2024 Sep 10. PMID 39270695